CLINICAL TRIAL: NCT01680692
Title: A Prospective, Randomized Study Comparing Continuous Femoral and Tibial Nerve Blocks vs. Continuous Femoral and Single Shot Sciatic Nerve Block in Total Knee Arthroplasties.
Brief Title: Continuous Femoral and Tibial Nerve Blocks in TKA Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Principal Investigator left institution--no subjects completed the study
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Collaborators: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E12094
Record Dates: First submitted 2012-08-29; First posted 2012-09-07 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Analgesia in Total Knee Arthroplasty
Keywords: Analgesia TKA; Total knee arthroplasty; Continuous femoral catheter; Continuous tibial catheter; Single shot sciatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous femoral and single shot sciatic nerve block (Active Comparator): Will receive pre-operative continuous femoral catheter & post-operative single shot sciatic with both given an initial bolus of 30 mL (femoral) 0.5% Ropivicaine & 20mL (sciatic) 0.2% Ropivicaine. Following surgery the femoral infusion will be started, which will be running Ropivicaine 0.2 at 10cc/hr.
  Interventions: Drug: Ropivicaine; Device: Continuous Femoral Nerve Catheter
- Continuous femoral and tibial peripheral nerve catheters (Experimental): Patients will receive pre-operative continuous femoral catheter & post-operative continuous tibial catheter with an initial bolus of 30 mL 0.5% Ropivicaine (femoral) & 20mL 0.2% Ropivicaine (tibial), which will be followed by infusions post-operatively running at 10cc/hr.
  Interventions: Drug: Ropivicaine; Device: Continuous Femoral Nerve Catheter; Device: Continuous Tibial Nerve Catheter

INTERVENTIONS:
Drug: Ropivicaine — Infusion of local anesthetic for post-operative analgesia.
Device: Continuous Femoral Nerve Catheter — Continuous femoral nerve catheter placed to deliver infusions of local anesthetic post-operatively.
  Other Names: Continous femoral nerve catheter infusion
Device: Continuous Tibial Nerve Catheter — Continuous infusion of local anesthetic delivered through a tibial nerve catheter post-operatively.
  Other Names: Continuous tibial nerve catheter infusion
  Arms: Continuous femoral and tibial peripheral nerve catheters

SUMMARY:
The purpose of this study is to evaluate whether a new regional anesthesia technique would provide better pain control, patient satisfaction, less narcotic use and no symptoms of foot drop after knee replacement surgery.

DETAILED DESCRIPTION:
The aim of this study is to compare and measure the effects of Ropivicaine given through catheters located in the femoral and tibial nerves on indices of sensory blockade after total knee arthroplasties. This is a randomized, prospective study designed to address the primary research question: Does placing a continuous femoral & tibial catheter infusion lead to superior analgesia and patient satisfaction during the entire hospital stay? The secondary research question is: Will selectively placing a continuous tibial catheter decrease the episodes of transient foot drop to zero? Investigators know from own regional institutional practices that by performing a continuous femoral with a single shot sciatic nerve block provides adequate analgesia of the entire leg, but by post-operative day 2 patient's begin to experience pain with rehabilitation and rest in the posterior-lateral aspect of the knee and leg secondary to wearing off of the sciatic nerve block anesthetic. Also, it is known that by blocking the sciatic nerve proximal to its bifurcation may lead to episodes of transient foot drop due to common peroneal nerve blockage and irritation. It is hypothesized that placement of continuous catheters in the femoral and tibial nerves would provide better analgesia and lead to no episodes of foot drop as compared to the patients that receive continuous femoral and single shot sciatic blocks.

Currently at Texas Tech Health Science Center-El Paso and University Medical Center, about 95% of patient's undergoing total knee arthroplasty's (TKAs) receives a continuous femoral infusion and a single shot sciatic with an initial bolus of 30mL (femoral) and 20mL (sciatic) of Ropivicaine 0.5% and an infusion of Ropivicaine 0.2% at a rate of 10cc/hr (usually started post-op) for at least the first 48-72 hours post-operatively. For our study, Orthopedic clinic will provide a copy of the consent form to the subject so that they can review it, and if interested in participating in the study, the patient can then contact the Principal Investigator or Study Coordinator directly. After informed consent is obtained, patients will be randomized during that time using a numbering system enclosed in sealed envelopes. Group 1 will receive a pre-operative continuous femoral catheter and a post-operative single shot sciatic with both given an initial bolus of 30 mL (femoral) 0.5% Ropivicaine and 20mL (sciatic) 0.2% Ropivicaine. Following surgery the femoral infusion will be started, which will be running Ropivicaine 0.2 at 10cc/hr. Group 2 will receive a pre-operative continuous femoral catheter and a post-operative continuous tibial catheter with an initial bolus of 30 mL 0.5% Ropivicaine (femoral) and 20mL 0.2% Ropivicaine (tibial), which will be followed by infusions post-operatively running at the same rate and dosage as group 1. All nerve blocks performed will be placed using a nerve stimulator (with no twitches lower than 0.2mA) under ultrasound-guidance. Proper catheter placement will be confirmed by injecting 3mL of air and visualizing by ultrasound. Once confirmed, the bolus dose as mentioned earlier of either Ropivicaine 0.5% (femoral) or 0.2% (sciatic/tibial) will be injected. All TKA cases will be performed under general anesthesia with laryngeal mask airway. Considering the fact that by placing a selective continuous tibial catheter pre-operatively, we run the risk of the catheter being the surgical field during the case. For this reason, it was decided that placement after the procedure would be best. Therefore, the patient will be taken back to the block room post-operatively and a continuous tibial nerve catheter or single shot (depending on what group assigned) will be placed and bolused using the same technique as previously described. To detect a 30% reduction in the pain score from 3-4 to a 1-2 would be required for an observed post-operative pain control difference. In order to achieve a statistically significant result to detect the previously observed difference, a sample of 38 patients in each group (total of 76) would be required. Assuming a high consent rate and given the fact many TKA's it is projected that this study can be completed in approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-85 years old) undergoing elective total knee arthroplasty's
* American Society of Anesthesiology Classification (ASA) 1, 2, or 3

Exclusion Criteria:

* Patient refusal

  * Under 18
  * Pregnancy
  * Presence of neurological disease or existing parasthesia
  * Diabetes
  * Chronic drug use
  * Infection of leg
  * American Society of Anesthesiology Classification (ASA) 4-6 (unstable conditions)
  * History of allergy to local anesthetics or opioids

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Post-Operative Analgesia | Patients pain score will be evaluated after surgery until discharge, an average of 3 to 4 days.
  Will measure pain using visual analog scale.

SECONDARY OUTCOMES:
Foot Drop | Evaluated in the first 24, 48, 72 hours prior to discharge.
  Daily lower extremity neurological examination of the foot (specifically dorsiflexion.

OTHER OUTCOMES:
Patient Satisfaction | Evaluated every 24, 48 and 72 hours prior to discharge.
  Patient satisfaction assessed using a daily numeric scale form (1-5 with 5 being most satisfied).
Opioid Consumption | Evaluated every 24, 48, 72 hours prior to discharge.
  Compare the total consumption of opioid use in study patients compared to control patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Teissler, MD, Principal Investigator — Texas Tech University Health Sciences Center- Paul L. Foster School of Medicine of El Paso; John Zaki, MD, Principal Investigator — Texas Tech University Health Sciences Center- Paul L. Foster School of Medicine of El Paso
Locations (1):
- University Medical Center of El Paso, Texas Tech University Health Sciences Center, El Paso, Texas, United States

REFERENCES:
- See also: Related Info — http://elpaso.ttuhsc.edu/som/anesthesiology/